CLINICAL TRIAL: NCT00293332
Title: A Phase II Study of Neoadjuvant Therapy With Docetaxel, Carboplatin, and Bevacizumab in Patients With Resectable Early Stage Non-Small Cell Lung Cancer
Brief Title: Docetaxel, Carboplatin, and Bevacizumab in Treating Patients With Stage I, Stage II, or Stage III Non-Small Cell Lung Cancer That Can Be Removed By Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to low subject accrual
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sarita Dubey, M.D., UCSF
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000455640; UCSF-04652; UCSF-IIT-12198; UCSF-H5535-25047-01A
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2007-06

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Carboplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: bevacizumab — Neoadjuvant therapy with 15 mg/kg, IV on Day 1 of each 21 day cycle for the first 2 cycles.
  Other Names: Avastin
Drug: carboplatin — Neoadjuvant therapy, AUC 6, IV on day 1 of each 21 day cycle for 3 cycles.
  Other Names: Paraplatin
Drug: docetaxel — Neoadjuvant therapy, 75 mg/m2, IV on day 1 of each 21 day cycle for 3 cycles.
  Other Names: Taxotere
Procedure: conventional surgery — Standard surgery after 3 cycles of neoadjuvant therapy with docetaxel, carboplatin, and bevacizumab. Bevacizumab is given for the first 2 cycles only.
  Other Names: Resection

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving docetaxel and carboplatin together with bevacizumab before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying how well giving docetaxel and carboplatin together with bevacizumab works in treating patients with stage I, stage II, or stage III non-small cell lung cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the clinical response rate in patients with stage IB-IIIA non-small cell lung cancer treated with neoadjuvant docetaxel, carboplatin, and bevacizumab.

Secondary

* Determine the median and overall survival of patients treated with this regimen.
* Determine the safety profile of this regimen.
* Determine the time to treatment failure of patients treated with this regimen.
* Determine the pathologic response rate and the resectability rate in patients treated with this regimen.
* Correlate vascular endothelial growth factor (VEGF) levels or expression with response and survival of patients treated with this regimen.

OUTLINE: Patients receive docetaxel IV over 15-60 minutes, carboplatin IV over 30-60 minutes, and bevacizumab* IV over 30-90 minutes on day 1. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Approximately 4-6 weeks after completion of chemotherapy, eligible patients with no distant or mediastinal disease progression undergo lobectomy, pneumonectomy, or segmentectomy with standard radical mediastinal lymph node dissection.

NOTE: *Bevacizumab is only administered during courses 1 and 2.

After completion of study treatment, patients are followed periodically for 8 years.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer

  * No squamous cell carcinoma
  * No histology in close proximity to a major vessel
* Resectable stage IB-IIIA disease
* No CNS or brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8.0 g/dL
* Bilirubin normal
* Creatinine ≤ 1.5 mg/dL
* Urine protein:creatinine < 1.0
* Alkaline phosphatase (AP), AST, and ALT must meet 1 of the following criteria:

  * AP normal AND AST and ALT ≤ 5 times upper limit of normal (ULN)
  * AP ≤ 2.5 times ULN AND AST and ALT ≤ 1.5 times ULN
  * AP ≤ 5 times ULN AND AST and ALT normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after completion of study treatment
* Adequate pulmonary and cardiovascular function to tolerate surgical resection
* No cavitation or history of hemoptysis (i.e., bright red blood ≥ ½ teaspoon)
* No existing peripheral neuropathy ≥ grade 1
* No known history of severe hypersensitivity reaction to drugs formulated with polysorbate 80
* No history of serious systemic disease, including any of the following:

  * Myocardial infarction within the past 6 months
  * Uncontrolled hypertension (i.e., blood pressure > 150/110 mm Hg on medication)
  * Unstable angina
  * New York Heart Association class II-IV congestive heart failure
  * Unstable symptomatic arrhythmia requiring medication

    * Patients with chronic atrial arrhythmia (i.e., atrial fibrillation or paroxysmal supraventricular tachycardia) are eligible
  * Clinically significant peripheral vascular disease (i.e., grade II or higher)
* No history of significant neurological or psychiatric condition
* No known active infection within the past 14 days
* No serious, nonhealing wound, ulcer, or bone fracture
* No evidence of bleeding diathesis or coagulopathy
* No stroke within the past 6 months
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
* No other serious illness or medical condition
* No active infection
* No other currently active malignancy except nonmelanoma skin cancer

  * Malignancies for which therapy has been completed and are considered to have ≤ 30% chance of risk of relapse are not considered active

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or VEGF inhibitor
* No prior (i.e., within the past 4 weeks), concurrent, or anticipated participation in another experimental drug study except a Genentech-sponsored bevacizumab cancer study
* No major surgical procedure, open biopsy, or significant traumatic injury within the past 28 days
* No anticipation for major surgical procedure during study treatment
* No fine-needle aspiration or core biopsy within 7 days prior to study entry
* No concurrent full-dose anticoagulation
* No other concurrent chemotherapy, immunotherapy, radiotherapy, or investigational therapy for this cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2005-12; Primary Completion 2007-03 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Clinical response rate by CT scan after 3 courses of induction treatment | After 3 cycles of induction treatment

SECONDARY OUTCOMES:
Pathologic response rate after 3 courses of induction treatment | After 3 cycles of induction treatment
Resectability rate after 3 courses of induction treatment | After 3 cycles of induction treatment
Median survival at 2 years after surgery | 2 years after surgery
Safety after 3 courses of induction treatment | After 3 cycles of induction treatment
Overall survival at 2 years after surgery | 2 years after surgery
Time to treatment failure within 2 years after surgery | 2 years after surgery
Correlation of serum VEGF levels prior to neoadjuvant therapy with primary and secondary objectives prior to start of induction treatment | Before induction treatment
Correlation of serum VEGF expression in resected tumor with primary and secondary objectives | After surgical removal of tumor
Correlation of VEGF levels measured immediately after resection and after adjuvant bevacizumab therapy with primary and secondary objectives | After resection and after adjuvant bevacizumab
Assay additional downstream VEGF activation pathway markers | At any time during the study

CONTACTS AND LOCATIONS:
Overall Officials: Sarita Dubey, MD, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Comprehensive Cancer Center, San Francisco, California, United States